CLINICAL TRIAL: NCT03655678
Title: A Phase 1/2/3 Study of the Safety and Efficacy of a Single Dose of Autologous CRISPR-Cas9 Modified CD34+ Human Hematopoietic Stem and Progenitor Cells (hHSPCs) in Subjects With Transfusion-Dependent β-Thalassemia
Brief Title: A Safety and Efficacy Study Evaluating CTX001 in Participants With Transfusion-Dependent β-Thalassemia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Collaborators: CRISPR Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTX001-111; 2024-516894-57-00 (Other: EU CT Number)
Record Dates: First submitted 2018-08-29; First posted 2018-08-31 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Beta-Thalassemia; Thalassemia; Genetic Diseases, Inborn; Hematologic Diseases; Hemoglobinopathies
Keywords: CRISPR-Cas9; Beta-Thalassemia; Hemoglobinopathies
MeSH Terms: conditions — beta-Thalassemia; Thalassemia; Genetic Diseases, Inborn; Hematologic Diseases; Hemoglobinopathies | interventions — exagamglogene autotemcel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- CTX001 (Experimental): CTX001 (autologous CD34+ hHSPCs modified with CRISPR-Cas9 at the erythroid lineage-specific enhancer of the BCL11A gene). Participants will receive a single infusion of CTX001 through a central venous catheter.
  Interventions: Biological: CTX001

INTERVENTIONS:
Biological: CTX001 — Administered by IV infusion following myeloablative conditioning with busulfan
  Other Names: Exagamglogene autotemcel; Exa-cel

SUMMARY:
This is a single-arm, open-label, multi-site, single-dose Phase 1/2/3 study in participans with transfusion-dependent β-thalassemia (TDT). The study will evaluate the safety and efficacy of autologous CRISPR-Cas9 Modified CD34+ Human Hematopoietic Stem and Progenitor Cells (hHSPCs) using CTX001.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosis of transfusion-dependent β-thalassemia (TDT) as defined by

  1. Documented homozygous β-thalassemia or compound heterozygous β-thalassemia including β-thalassemia/hemoglobin E (HbE). Participants can be enrolled based on historical data, but a confirmation of the genotype using the study central laboratory will be required before busulfan conditioning
  2. History of at least 100 mL/kg/year or ≥10 units/year of packed RBC transfusions in the prior 2 years before signing the consent or the last rescreening for patients going through re-screening
* Eligible for autologous stem cell transplant as per investigator's judgment

Key Exclusion Criteria:

* A willing and healthy 10/10 Human Leukocyte Antigen (HLA)-matched related donor is available per investigator's judgement
* Prior allo-HSCT
* Participants with associated α-thalassemia and >1 alpha deletion or alpha multiplications
* Participants with sickle cell beta thalassemia variant
* Clinically significant and active bacterial, viral, fungal, or parasitic infection as determined by the investigator
* White blood cell (WBC) count <3 × 10^9/L or platelet count <50 × 10^9/L not related to hypersplenism

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 59 (Actual)
Dates: Start 2018-09-14 (Actual); Primary Completion 2025-11-13 (Actual); Study Completion 2025-11-13 (Actual)

PRIMARY OUTCOMES:
Proportion of participants achieving transfusion independence for at least 12 consecutive months (TI12) | From 60 days after last RBC transfusion up to 24 months post-CTX001 infusion]
Proportion of participants with engraftment (first day of 3 consecutive measurements of absolute neutrophil count [ANC] ≥500/µL on three different days) | Within 42 days after CTX001 infusion
Time to neutrophil and platelet engraftment | Days post-infusion to engraftment
Frequency and severity of collected adverse events (AEs) | Signing of informed consent through Month 24 visit
Incidence of transplant-related mortality (TRM) | Baseline (pre-transfusion) to 100 days and 1 year post-CTX001 infusion
All-cause mortality | Signing of informed consent through Month 24 visit

SECONDARY OUTCOMES:
Proportion of participants achieving transfusion independence for at least 6 consecutive months (TI6) | From 60 days after last RBC transfusion up to 24 months post-CTX001 infusion
Proportion of participants achieving at least 95 percent (%), 90%, 85%, 75%, and 50% reduction from baseline in annualized volume of RBC transfusions after Month 10 after CTX001 infusion | From Month 10 up to 24 months post-CTX001 infusion
Relative reduction from baseline in annualized volume of RBC transfusions after Month 10 after CTX001 infusion | From Month 10 up to 24 months post-CTX001 infusion
Duration of transfusion free in participants who have achieved TI12 | From 60 days after last RBC transfusion up to 24 months post-CTX001 infusion
Proportion of alleles with intended genetic modification in peripheral blood leukocytes over time | Day 1 CTX001 infusion through Month 24 visit
Proportion of alleles with intended genetic modification present in CD34+ cells of bone marrow over time | Day 1 CTX001 infusion through Month 24 visit
Change in fetal hemoglobin concentration over time | Baseline (pre-transfusion) through Month 24 visit
Change in total hemoglobin concentration over time | Baseline (pre-transfusion) through Month 24 visit
Change in health-related quality of life (HRQoL) from baseline over time using EuroQol Questionnaire (5 dimensions - 5 levels of severity - EQ-5D-5L) | Screening visit through Month 24 visit
  The EQ-5D-5L Questionnaire consists of the EQ-5D descriptive system and the EQ visual analogue scale (VAS). The EQ-5D comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort, anxiety/depression, and 5 levels: no problems to extreme problems. The subject marks the most appropriate statement in each dimension, resulting in a 1-digit number for that dimension. The digits can be combined in a 5-digit number describing the subject's health state. The EQ VAS records the subject's self-rated health on a 100-point VAS, endpoints labelled "the best health you can imagine" and "the worst health you can imagine."
Change in health-related quality of life (HRQoL) from baseline over time using the Functional assessment of cancer therapy-bone marrow transplant questionnaire (FACT-BMT) | Screening visit through Month 24 visit
  The FACT-BMT Questionnaire includes physical, social, family, emotional, and functional well-being, and treatment specific concerns of bone marrow transplantation. Each statement has a 5-point Likert-type response scale ranging from 0=not at all to 4=very much. The subject marks one number per line as it applies to the past 7 days. Questionnaires are scored; the higher the score, the better the QOL.
Change in patient reported outcome (PRO) over time assessed using EQ-5D-Youth (EQ-5D-Y) | Screening visit through Month 24 visit
Change in PRO over time assessed using pediatric quality of life inventory (PedsQL) | Screening visit through Month 24 visit
Changes in liver iron concentration (LIC) and cardiac iron content (CIC) and ferritin parameters of iron overload | Screening visit through Month 24 visit
Proportion of participants receiving iron chelation therapy | 1 month post-CTX001 infusion through Month 24 visit

CONTACTS AND LOCATIONS:
Locations (14):
- United States (6):
  - Lucile Packard Children's Hospital, Palo Alto, California
  - Ann & Robert Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Columbia University Medical Center (21+ years), New York, New York
  - Columbia University Medical Center, New York, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - The Children's Hospital at TriStar Centennial Medical Center/ Sarah Cannon Center for Blood Cancers, Nashville, Tennessee
- Canada (2):
  - The Hospital for Sick Children, Toronto
  - British Columbia Children's Hospital, Vancouver
- Germany (3):
  - Universitätsklinikum Düsseldorf Hospital Duesseldorf, Düsseldorf
  - Regensburg University Hospital, Clinic and Polyclinic for Paediatric and Adolescent Medicine, Regensburg
  - University Hospital Tübingen, Tübingen
- Ospedale Pediatrico Bambino Gesù, IRCCS, Rome, Italy
- United Kingdom (2):
  - Imperial College Healthcare NHS Trust, Hammersmith Hospital, London
  - University College London Hospitals NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/our-science/clinical-trials-data-sharing/

REFERENCES:
- [Derived] Fuente J, Frangoul H, Lang P, Wall D, Meisel R, Corbacioglu S, Li AM, Shah AJ, Carpenter B, Kwiatkowski JL, Mapara MY, Liem RI, Rupprecht J, Kuo KHM, Merkeley H, Algeri M, Smith W, Kohli P, Li N, Rubin J, Zhang S, Hobbs W, Locatelli F. Improvements in health-related quality of life in patients with transfusion-dependent beta-thalassemia after exagamglogene autotemcel. Blood Adv. 2025 Dec 23;9(24):6502-6510. doi: 10.1182/bloodadvances.2025016702. PMID 40862696
- [Derived] Locatelli F, Lang P, Wall D, Meisel R, Corbacioglu S, Li AM, de la Fuente J, Shah AJ, Carpenter B, Kwiatkowski JL, Mapara M, Liem RI, Cappellini MD, Algeri M, Kattamis A, Sheth S, Grupp S, Handgretinger R, Kohli P, Shi D, Ross L, Bobruff Y, Simard C, Zhang L, Morrow PK, Hobbs WE, Frangoul H; CLIMB THAL-111 Study Group. Exagamglogene Autotemcel for Transfusion-Dependent beta-Thalassemia. N Engl J Med. 2024 May 9;390(18):1663-1676. doi: 10.1056/NEJMoa2309673. Epub 2024 Apr 24. PMID 38657265
- [Derived] Brusson M, Miccio A. Genome editing approaches to beta-hemoglobinopathies. Prog Mol Biol Transl Sci. 2021;182:153-183. doi: 10.1016/bs.pmbts.2021.01.025. Epub 2021 Mar 1. PMID 34175041
- [Derived] Frangoul H, Altshuler D, Cappellini MD, Chen YS, Domm J, Eustace BK, Foell J, de la Fuente J, Grupp S, Handgretinger R, Ho TW, Kattamis A, Kernytsky A, Lekstrom-Himes J, Li AM, Locatelli F, Mapara MY, de Montalembert M, Rondelli D, Sharma A, Sheth S, Soni S, Steinberg MH, Wall D, Yen A, Corbacioglu S. CRISPR-Cas9 Gene Editing for Sickle Cell Disease and beta-Thalassemia. N Engl J Med. 2021 Jan 21;384(3):252-260. doi: 10.1056/NEJMoa2031054. Epub 2020 Dec 5. PMID 33283989